CLINICAL TRIAL: NCT00091494
Title: Socioeconomic Patterning of Inflammation and Hemostasis - Ancillary to MESA
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1268; R01HL076831 (NIH)
Record Dates: First submitted 2004-09-09; First posted 2004-09-13 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2008-07

CONDITIONS: Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Inflammation; Blood Coagulation Disorders
MeSH Terms: conditions — Atherosclerosis; Cardiovascular Diseases; Heart Diseases; Inflammation; Blood Coagulation Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To investigate how inflammation, hemostasis, and stress may contribute to neighborhood and individual-level socioeconomic differences in cardiovascular risk.

DETAILED DESCRIPTION:
BACKGROUND:

In epidemiologic studies, associations of cardiovascular risk with individual and neighborhood socioeconomic characteristics tend to persist after adjustment for established cardiovascular risk factors suggesting that other mediators may be involved. However, evidence regarding what these mediators may be is largely absent. Elucidating the reasons for these persistent socioeconomic differences may enhance our ability to reduce these differentials and will contribute to our understanding of the causes of cardiovascular disease generally. Two biological processes, inflammation and hemostasis, have recently emerged as potentially important in the development of atherosclerosis and the precipitation of clinical cardiovascular events. Both processes have also been recently linked to psychosocial factors and stress. However, studies investigating social gradients in inflammation and hemostasis remain rare. In addition, the relation of psychosocial factors and biological markers of the stress response to inflammation and hemostasis have not been examined in large population-based studies.

DESIGN NARRATIVE:

The study is ancillary to the ongoing epidemiologic study of atherosclerosis, the Multi-Ethnic Study of Atherosclerosis (MESA). The project will collect data on stress hormones and follow- up measures of inflammation and hemostasis which are not part of the existing MESA protocol on a subsample of the cohort. The study will also collect additional data on neighborhood sources of stress for the subsample. The new data will be linked to existing MESA data.

Using newly collected data linked to the MESA, the study will investigate (1) associations of neighborhood and individual-level socioeconomic indicators with markers of inflammation and hemostasis; (2) associations of individual-level psychosocial factors and sources of chronic stress (at the individual and neighborhood level) with inflammatory markers and hemostasis; and (3) the relationship between biological markers of the stress response (such as cortisol and adrenaline/noradrenaline) and inflammation and hemostasis). Project aims will be achieved by linking MESA data to newly-collected data on neighborhood characteristics and biomarkers of inflammation, hemostasis and the stress response in MESA participants. The project is innovative in that it will span and link three levels: the social/environmental level (neighborhood characteristics and social position), the behavioral/psychological level (behavioral and psychosocial factors), and the biological level (inflammation, hemostasis, and stress hormones). The study will provide a unique opportunity to elucidate the links between socioeconomic factors, stress, inflammation and hemostasis in a large and diverse population-based sample.

ELIGIBILITY:
Participants at NY and LA MESA sites.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an ancillary study to MESA.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2004-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Diez Roux, Principal Investigator — University of Michigan